CLINICAL TRIAL: NCT01232205
Title: Antioxidant Supplementation in Pregnant Women With Low Antioxidant Status
Brief Title: Antioxidant Supplementation in Pregnant Women
Acronym: ASIP1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Showa University (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Yuditiya Purwosunu, Dept Obstetrics Gynecology, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: asip02
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Pregnant Women; Preeclampsia
Keywords: antioxidant supplementation; preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- micronutrient antioxidant (Active Comparator): Supplementation with milk enriched with vitamin and mineral, such as Cu, Zn, Mn, Fe, carotene, vitamin B6, B12, C, E, selenium, and calcium
  Interventions: Dietary Supplement: micronutrient antioxidant
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: micronutrient antioxidant — Supplementation with milk enriched with vitamin and mineral, such as Cu, Zn, Mn, Fe, carotene, vitamin B6, B12, C, E, selenium, and calcium
  Other Names: antioxidant
  Arms: micronutrient antioxidant
Dietary Supplement: Control — supplementation with milk
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the benefit of several micro nutrients of antioxidants (using milk) in a cohort of women with low antioxidant status and the changes in cell-free mRNA.

DETAILED DESCRIPTION:
Preeclampsia remains one of leading causes of maternal and perinatal mortality and morbidity. Despite intensive research, the cause of preeclampsia has not been established. One of the theories is exaggeration of systemic inflammatory that might induce reactive oxygen species (ROS). It has been proposed that pregnancy will progress uneventfully if adequate antioxidant exists to buffer ROS. The ROS can induce endothelial dysfunction which leads to clinical symptoms of hypertension and proteinuria in preeclampsia. Several large randomized clinical trials of antioxidant supplementation have concluded that there were no benefits of antioxidants supplementation for prevention of preeclampsia. However, there is limited information about benefits of antioxidants in women with low antioxidant status at early gestation that deprived of the antioxidant most. Our aim, therefore, in this study was to assess whether early supplementation with milk enriched with vitamin and mineral, such as Cu, Zn, Mn, Fe, carotene, vitamin B6, B12, C, E, selenium, and calcium lowers the risk of preeclampsia in women with low antioxidant status at early gestation.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with 8-12 weeks of gestation

Exclusion Criteria:

* known multiple pregnancy
* known fetal anomaly
* known thrombophilia
* known infections and mola hydatidosa
* chronic renal failure
* uncontrolled hypertension
* known placental abnormalities
* documented uterine bleeding within a week of screening
* uterine malformation
* history of medical and metabolic complication such as heart disease or diabetes

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2001-06; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noroyono Wibowo, MD, PhD, Study Director — Dept Obstetrics Gynecology, Indonesia University; Yuditiya Purwosunu, MD, Principal Investigator — Dept Obstetrics Gynecology Indonesia University
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Derived] Wibowo N, Purwosunu Y, Sekizawa A, Farina A, Idriansyah L, Fitriana I. Antioxidant supplementation in pregnant women with low antioxidant status. J Obstet Gynaecol Res. 2012 Sep;38(9):1152-61. doi: 10.1111/j.1447-0756.2012.01855.x. Epub 2012 May 8. PMID 22563751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in June 2001 and completed in December 2009, Department of Obstetrics and Gynaecology, University of Indonesia, at Cipto Mangunkusumo National Hospital
Pre-assignment Details: There were 110 (65.4 percent) eligible subjects from 168 pregnant women, because of ferric reducing ability of plasma (FRAP) level measured
Period: Overall Study
Arm/Group | Micronutrient Antioxidant | Control
Started | 52 | 58
Completed | 49 | 55
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micronutrient Antioxidant | Control | Total
Number analyzed (Participants) | 52 | 58 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 58 | 110
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.1 (5.08) | 29.7 (5.07) | 28.9 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 58 | 110
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Indonesia | 52 | 58 | 110

OUTCOME MEASURES:

1. Primary Outcome: Preeclampsia
Description: Preeclampsia was defined as gestational hypertension (systolic pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg [Korotkoff V] on ≥ 2 occasions after 20 weeks gestation) with proteinuria (> 0.3 g/day). Severe preeclampsia was defined by the presence of >1 of the following: (a) severe gestational hypertension (systolic pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg on 2 occasions after gestational week 20), or (b) severe proteinuria (≥5g protein in a 24-h urine specimen or ≥3 g in 2 random urine samples collected ≥4 h apart)
Time Frame: 40 weeks
Reporting Status: Not Posted

2. Secondary Outcome: Cell-free mRNA
Description: Secondary outcome were level of mRNA level of angiogenic factors (vascular endothelial growth factor receptor-1 (VEGFR-1), placental growth factor (PlGF) and endoglin(ENG)); antioxidant status (FRAP, heme oksigenase-1 (HO-1) and superoxide-dismutase (SOD))
Time Frame: 40 weeks
Reporting Status: Not Posted

3. Primary Outcome: Preeclampsia
Description: as for outcome 1
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | Micronutrient Antioxidant | Control
Number analyzed (Participants) | 52 | 58
participants | 1 | 8

ADVERSE EVENTS:
Time Frame: nine months
Description: monthly questionare
Arm/Group | Micronutrient Antioxidant | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No